CLINICAL TRIAL: NCT04008108
Title: A Pilot Study to Evaluate the Variation of Physical Activity, Measured by the Number of Steps Per Day, After Artificial Urinary Sphincter Implantation
Brief Title: Variation of Physical Activity, Measured by the Number of Steps Per Day, After Artificial Urinary Sphincter Implantation
Acronym: AP-SU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP190234; 2019-A00680-57 (Other: ANSM)
Record Dates: First submitted 2019-04-15; First posted 2019-07-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; artificial urinary sphincter; physical activity; number of steps per day; activity tracker
MeSH Terms: conditions — Urinary Incontinence; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with urinary incontinence (Experimental): Patient with urinary incontinence
  Interventions: Other: Activity sensor

INTERVENTIONS:
Other: Activity sensor — Activity sensor worn on the wrist during 7 days, 24h/24 to evaluate physical activity of patient (measured by the number of step per day) before and after Artificial Urinary Sphincter Implantation.

SUMMARY:
The management of urinary incontinence seems to improve daily activities and the practice of physical activity, according to the literature. Unfortunately, all of these studies are based on self-questionnaires with the disadvantages of self-evaluation, more subjective.

For several years activity sensors have been used in the medical field (rheumatology, cardiology, diabetology, etc.). They allowed the evaluation of physical activity in real life situations, whether to evaluate the degree of severity of a pathology or the impact of a new treatment on the resumption of activities.

Activity sensors are devices that transform body motion into digital measurements. They provide detailed information on the frequency, duration, intensity and type of movement to determine, for example, the number of steps taken, the distance traveled, calories burned and the quality of sleep.

It is hypothesized that urinary incontinence treatment can increase physical activity and so improve the quality of life of patients, that can be measure by activity sensors.

DETAILED DESCRIPTION:
The management of urinary incontinence seems to improve daily activities and the practice of physical activity, according to the literature. Unfortunately, all of these studies are based on self-questionnaires with the disadvantages of self-evaluation, more subjective.

The artificial urinary sphincter (AUS) implantation is an effective treatment on stress urinary incontinence in men and women. Currently the PadTest/24 hours is the reference for his evaluation.

For several years activity sensors have been used in the medical field (rheumatology, cardiology, diabetology, etc.). They allowed the evaluation of physical activity in real life situations, whether to evaluate the degree of severity of a pathology or the impact of a new treatment on the resumption of activities.

Activity sensors are devices that transform body motion into digital measurements. They provide detailed information on the frequency, duration, intensity and type of movement to determine, for example, the number of steps taken, the distance traveled, calories burned and the quality of sleep.

It is hypothesized that urinary incontinence treatment can increase physical activity and so improve the quality of life of patients, that can be measure by activity sensors.

The research is a monocentric, prospective study.

The Primary objective of this study is to evaluate the variation of physical activity measured by the number of steps per day, before AUS implantation and 3 months after the activation of the sphincter.

For that, the primary outcome measure is the number of steps per day measured 24h/24 for 7 consecutive days by activity sensor, before AUS implantation and 3 months after activation of the sphincter.

All adult patients (men and women) with a surgical indication for urinary incontinence treatment by AUS in the urology department of Pitié-Salpêtrière hospital will be screened for eligibility.

Four visits will be programed as standard of care :

* During the first visit, patients will be informed of the study and their agreement will be recorded. Patients' eligibility will be checked.
* AUS implantation
* AUS activation
* AUS follow-up, around fourteen weeks after activation The activity sensor, the Pad/Test/24 hours and questionnaires such as eQOL will be performed at home before AUS implantation, 1 month after the AUS activation and 3 months after the AUS activation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Surgical indication of urinary incontinence treatment with artificial urinary sphincter implantation
* Patient informed and not opposed to the research
* Reading and speaking comprehension of the French language

Exclusion Criteria:

* Patient under guardianship or curators
* Contraindication to the placement of an artificial urinary sphincter
* Patients requiring walking assistance (canes, walker, wheelchair)
* Revisions of artificial urinary sphincter already implanted
* Cognitive impairment deemed incompatible with research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Number of steps per day, during 7 days at 3 months of the AUS activation | Through the study completion, an average of 8 months
  Number of steps per day measured 24h/24 for 7 consecutive days by the activity sensor, at 3 months after activation of the AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).

SECONDARY OUTCOMES:
Number of steps per day, during 7 days, at 1 month of the AUS activation | Through the study completion, an average of 6 months
  Number of steps per day measured 24h/24 for 7 consecutive days by the activity sensor, at 1 month after activation of the AUS.
  1 month after activation of the AUS is corresponding to 24 weeks from the inclusion (6 months).
Other activity sensor data (heart rate) | Through the study completion, an average of 8 months
  Heart rate measured by the activity sensor preoperatively and at 1 month and 3 months after activation of the AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).
Other activity sensor data (sedentary and activity percentage in the day) | Through the study completion, an average of 8 months
  Sedentary and activity percentage a day measured by the activity sensor preoperatively and at 1 month and 3 months after activation of the AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).
Incontinence Quality of Life (I-QOL) | Through the study completion, an average of 8 months
  I-QOL is a self-report Quality of Life measure specific to urinary problems. The I-QOL is commonly used and consists of 22 items, all of which use a five-point ordinal response scale in which 1 = extremely, 2 = quite a bit, 3 = moderately, 4 = a little, and 5 = not at all.
  I-QOL scores are transformed to a 0-100 scale for easy interpretability. Higher scores indicate better quality of life.
  Scale score = ((The sum of the items - lowest possible score) / Possible raw score range ) x 100.
  Questionnaire I-QoL fulfilled before implantation and 3 months after activation of AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).
International Physical Activity Questionnaire (IPAQ) | Through the study completion, an average of 8 months
  IPAQ is a 8 items questionnaire that assess 3 types of activity (walking, moderate-intensity activities and vigorous-intensity activities) in the following domains: leisure time, domestic/gardening, work-related, transport-related. It provide separate scores on each type of activity. Computation of the total score requires summation of the duration (in minutes) and frequency (days) of each type of activity. A Metabolic Equivalent Task (MET) is a multiple of the estimated resting energy expenditure.
  Walking MET-minutes/week=3.3*walking minutes*walking days Moderate MET-minutes/week=4.0*moderate-intensity activity minutes*moderate days Vigorous MET-minutes/week=8.0*vigorous-intensity activity minutes*vigorous-intensity days Total =sum of Walking+Moderate+Vigorous METminutes/week scores.
  Questionnaire IPAQ fulfilled before implantation and 3 months after activation of AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).
PAD-test / 24h | Through the study completion, an average of 8 months
  PAD-test / 24h performed at home preoperatively and 3 months after activation of AUS.
  3 months after activation of the AUS is corresponding to 32 weeks from the inclusion (8 months).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MOZER, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service d'Urologie, Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No